CLINICAL TRIAL: NCT04832594
Title: Image Analysis With Artificial Intelligence to Increase Precision in Breast Cancer Screening - the ScreenTrust MRI Substudy: a Prospective Trial of AI to Select Women for Supplemental Screening MRI
Brief Title: Using AI to Select Women for Supplemental MRI in Breast Cancer Screening
Acronym: ScreenTrustMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: KTH Royal Institute of Technology (Other); Region Stockholm (Other Government); Bröstcancerförbundet, Sweden (Unknown)
Responsible Party: Principal Investigator, Fredrik Strand, Principal Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KSRAD001
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Artificial Intelligence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: For each screening mammography examination, the AI tool will produce an AI Joint Score and an AI Masking Score. Women having an AI Masking Score above the threshold and an AI Joint Score above the threshold will be invited to the study unless they met exclusion criteria. Women who decide to participate, will be randomized to MRI or no-MRI (standard-of-care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemental MRI (Experimental): Women randomized to MRI will be examined using a shortened MRI protocol on a Signa Premier 3T MRI scanner. The MRI examination will be reviewed by two radiologists and assigned BI-RADS score. Appropriate clinical work-up will follow according to the BI-RADS score. BI-RADS 3 or higher at initial MRI will be recalled for a second look ultrasound.
  Interventions: Other: AI selection for supplemental breast MRI
- No MRI (standard-of-care) (No Intervention): Standard-of-care. Both arms will have had a regular screening mammography examination prior to randomization. The "No MRI" arm will have no further intervention.

INTERVENTIONS:
Other: AI selection for supplemental breast MRI — An AI tool will generate scores used to determine eligibility. Women randomized to MRI will be examined in an MRI scanner.
  Arms: Supplemental MRI

SUMMARY:
This is a prospective clinical trial aiming to determine the ability of an AI pipeline to identify women who would benefit from supplemental MRI in terms of decreasing the number of cancers having a significantly delayed detection

DETAILED DESCRIPTION:
All women attending mammography screening at Karolinska University Hospital will have their mammograms analyzed by AI (Figure 1). The specific AI-implementation (AI tool) in this study is a result of AI predictions from three equally weighted component AI models analyzing mammograms: (i) masking predictor, (ii) risk predictor and (iii) cancer signs predictor (by one commercial CAD model and one in-house academic CAD model); the age of the woman is also taken into account by multiplying the score with (110-age)/70. The purpose of the age factor is to attain a relatively similar proportion of MRI exams in the lower and higher age groups. The aim of the AI tool is to identify women with the highest probability of having a delay in cancer detection, i.e., having had a false negative screening mammogram.

An AI-based framework has been developed by researchers at Karolinska Institute (led by Dr. Fredrik Strand) and Royal Institute of Technology (led by Dr: Kevin Smith). The specific AI-implementation (AI tool) in this study is a result of AI predictions from three equally weighted component AI models analyzing mammograms: (i) masking predictor, (ii) risk predictor and (iii) cancer signs predictor (by one commercial CAD model and one in-house academic CAD model); the age of the woman is also taken into account by multiplying the score with (110-age)/70. The purpose of the age factor is to attain a relatively similar proportion of MRI exams in the lower and higher age groups. The aim of the AI tool is to identify women with the highest probability of having a delay in cancer detection, i.e., having had a false negative screening mammogram. The specific AI tool and its settings will remain the same during the study. For each examination, the AI tool will produce an AI Joint Score and an AI Masking Score. The AI Masking Score cut-off point was defined by the median of examinations collected during the initial period of March 1 to March 24, 2021. The cut-off point of the AI Joint Score was defined by the 92nd percentile of the initial population. Women meeting these criteria will be invited to the study, and randomized to MRI or no-MRI (standard-of-care).

A Signa Premier 3T MRI scanner from GE Healthcare will be used. The MRI protocol will contain a T2-weighted Dixon sequence and a T1-weighted dynamic contrast enhanced series, and will remain the same through the course of the study. All MRI exams will be assessed by two radiologists, where the second reader will have access to the assessment of the first reader. In case of disagreement, a consensus discussion between two radiologists will be held. The MRI exams will be assessed according to BI-RADS, and follow-up will depend on the BI-RADS category (Figure 2). Women with BI-RADS 1-2 will have no further diagnostics and will be sent a 'healthy letter'. Women with BI-RADS 3 to 5 will be recalled for 2nd look ultrasound. Women with BI-RADS 4-5 will be included in the regular process for established cancer suspicion and be discussed in a multidisciplinary team conference. For women with BI-RADS 3, the follow-up will be handled within the breast radiology unit.

ELIGIBILITY:
Inclusion Criteria:

* Complete four-view screening mammography examination

Exclusion Criteria:

* Women in surveillance program referred from the hereditary cancer unit
* Breast implants
* Prior breast cancer
* Breast feeding
* MRI contraindication requiring radiologist assessment
* AI Tool unable to process mammograms due to technical reason

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Significantly Delayed Breast Cancer Detection per 1000 women | Until 27 months from study inclusion (includes cancer detected at subsequent screening within this time frame). Cancer detected at the initial screening mammography or MRI shall not be included.
  Composite end-point defined by either: 1. Interval Cancer, 2. Cancer with lymph node metastasis, 3. Cancer with invasive component larger than 15 mm

SECONDARY OUTCOMES:
MRI-detected breast cancer | Diagnosis during work-up within 2 months of the initial screening MRI
  Breast cancer detected at the initial screening MRI for women in the Intervention arm of the study
Invasiveness | All diagnosed breast cancer within 27 months of study inclusion
  In situ and/or Invasive cancer
Histology | All diagnosed breast cancer within 27 months of study inclusion
  Ductal, Lobular, Mucinous, Tubular, Other
Lymph node metastasis | All diagnosed breast cancer within 27 months of study inclusion
  0 nodes, 1-3 nodes, 4 or more nodes
Tumor size | All diagnosed breast cancer within 27 months of study inclusion
  Size (in millimetre) for the invasive and the in situ component
Receptor status | All diagnosed breast cancer within 27 months of study inclusion
  ER positive/negative, PR positive/negative, HER2 positive/negative
Age | At study inclusion
  Age of the woman
Distribution of AI scores | At study inclusion
  Histogram, mean, median and dispersion measures for the AI Scores
BI-RADS codes | At study inclusion and until end of 27 month follow-up
  For each MRI examination, the BI-RADS code for fibroglandular volume, background enhancement and breast lesions
Biopsy result | Diagnosis during work-up within 2 months of the MRI examination
  Pathology assessment of biopsy: normal tissue, benign lesion, cancer in situ, invasive cancer
Participant questionnaire | At study inclusion
  Participant questionnaire replies for MRI contraindications and for Breast cancer-related history

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Strand, MDPhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The final trial dataset will be available for the research team of the principal investigator. Pseudonymized data can be made available for external research audit. Anonymous data may be shared with academic researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available during study time and until 2 years after publication of any manuscript resulting from the study
Access Criteria: Data Transfer Agreement must be signed. Request must be made by an academic researcher at an internationally recognized university.

REFERENCES:
- [Derived] Salim M, Liu Y, Sorkhei M, Ntoula D, Foukakis T, Fredriksson I, Wang Y, Eklund M, Azizpour H, Smith K, Strand F. AI-based selection of individuals for supplemental MRI in population-based breast cancer screening: the randomized ScreenTrustMRI trial. Nat Med. 2024 Sep;30(9):2623-2630. doi: 10.1038/s41591-024-03093-5. Epub 2024 Jul 8. PMID 38977914

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04832594/Prot_SAP_001.pdf